CLINICAL TRIAL: NCT07173049
Title: Speech Supplementation Strategies for Improving Intelligibility in Children With Cerebral Palsy (CP)
Brief Title: Speech Production Enhancement Using Augmentative Communication for Kids
Acronym: SPEAK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0885; 2R01DC009411-16 (NIH); A481800 (Other: UW Madison); L&S/COMMUN SCI & DISORDERS (Other: UW Madison); Protocol Version 7/21/2025 (Other: UW Madison)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP); Intelligibility, Speech; Augmentative and Alternative Communication
Keywords: Cerebral Palsy; Speech; Intelligibility; Speech supplementation; Augmentative and alternative communication
MeSH Terms: conditions — Cerebral Palsy; Speech Intelligibility; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- speech supplementation (Experimental): Children will complete a pre-test on their speech prior to learning speech supplementation strategy use, and will be taught to use speech supplementation through one-on-one teaching. They will then complete a post test on their speech while using speech supplementation.
  Interventions: Behavioral: AAC Speech supplementation

INTERVENTIONS:
Behavioral: AAC Speech supplementation — The speech supplementation intervention involves learning to point to pictures, words, or letters on a communication board while simultaneously producing speech. Children will spend up to 30 minutes learning to use the strategy in one- on-one interaction with a speech therapist and demonstrate mastery by using the strategy successfully on a series of test stimuli.

SUMMARY:
The goal of this clinical trial is to learn if speech supplementation can improve speech intelligibility in children ages 7 to 17 years with cerebral palsy. The main questions it aims to answer are:

* To what extent can speech supplementation improve intelligibility in children with CP compared with habitual speech produced without speech supplementation?
* How much intelligibility change is necessary for meaningful improvement when children use speech supplementation strategies?

Participants will:

* complete speech and language assessments
* complete a speech pre-test using habitual speech
* learn a speech supplementation strategy with training from a speech-language pathologist
* complete a speech post-test using the speech supplementation strategy

DETAILED DESCRIPTION:
This study uses a pre-/post- test design to test the effects of a one-session intervention to improve speech intelligibility in 100 children with cerebral palsy and dysarthria. The intervention involves the augmentative and alternative communication (AAC) strategy known as speech supplementation. Specifically, children will learn how to simultaneously speak and point to the first letter of each word on a communication board, or to speak and point to a topical picture on a communication board. The strategy serves to provide listeners with context cues for spoken words, and it also serves to impact temporo-acoustic features of speech by reducing rate of speech and making word boundaries clear.

In this study, children will first participate in a set of baseline assessment measures, which will include the production of a corpus of 60 sentences (referred to as "habitual speech"). Then, children will learn to use the speech supplementation strategy through one-on-one clinician modeling, teaching, and practice. When children have mastered the strategy on a set of practice sentences, they will complete a post-test in which they produce the same set of elicited sentences a second time using speech supplementation.

Pre-test and post-test speech samples will then be played to two groups of listeners. One group will orthographically transcribe the words produced by children in both conditions (habitual and supplemented). Listener transcriptions in each condition will be scored as correct or incorrect based on whether they matched the intended word. Average percent of words identified correctly will be obtained from 2 listener for each child and each speaking condition as measures of speech intelligibility. The difference between habitual speech (pre-test) and supplemented speech (post-test) will be examined to quantify the effects of the speech supplementation on intelligibility.

The second set of listeners will hear the same speech samples as the first set (habitual speech and supplemented speech), but they will make ratings of whether one of the conditions seems more understandable than the other, and if so, they will rate how much better using a 7-point Likert scale.

These two sets of data from listeners will enable us to measure the minimum detectable difference in speech intelligibility and then the minimal clinically important difference based on listener ratings. Together these measures will enable us to determine how much change in intelligibility is necessary in order for clinically meaningful improvement. The hypotheses are as follows:

1. speech supplementation will result in increased speech intelligibility relative to habitual speech.
2. the minimal clinically important difference in intelligibility scores to consider the speech supplementation strategy "successful" will vary depending on child severity, with more severely speech impaired children requiring a larger improvement to achieve a clinically meaningful change.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of cerebral palsy, or a similar, related condition that affects early motor development and presents as a chronic motor disability
* Age between 7 and 17 years
* Clinical dysarthria with speech intelligibility between 10-85 percent
* Able to produce connected speech in English, with a minimum utterance length of 3 words
* Able to use hands to point to items on a communication board
* Cognitive/language skills that enable basic picture identification on a communication board
* Pass pure tone hearing screening

Exclusion Criteria:

* Failure to meet all inclusion criteria.
* Vision impairment that precludes being able to see items on a communication board.
* Not suitable for participation due to other reasons at the discretion of the investigators.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Change in speech intelligibility scores from pre- to post- intervention as measured by listener transcription of speech samples | Before and after intervention within one session in a single day 1
  Quantify the change in speech intelligibility associated with the use of speech supplementation strategies by having listeners orthographically transcribe speech samples. Intelligibility scores are percentage calculations of the number of words identified correctly by listeners, ranging from 0 to 100 percent. Higher percentages reflect greater intelligibility, or a better understanding of what the speaker said by naive listeners.

SECONDARY OUTCOMES:
Perceived change in intelligibility from pre- to post-intervention as measured by listener ratings of the magnitude of difference between pre- and post- intervention speech samples. | Before and after intervention within one session in a single day 1
  Listener ratings of their perception of the magnitude of change in intelligibility between pre- and post-test speaking conditions. Listeners will hear pre- and post-intervention speech samples and will indicate whether they can hear a differences and if so, how large the differences was using a 5-point likert rating scale. Higher values on the scale reflect larger perceived differences.

OTHER OUTCOMES:
Exploratory: Change in speech rate from pre- to post- intervention as measured by difference in words per minute produced between pre- and post- intervention speech samples | Before and after intervention within one session in a single day 1
  The duration of each utterance produced, inclusive of pauses, will be measured as the total time between the onset of the first word and the offset of the last word. The number of words in each utterance will be divided by the utterance duration, which will be averaged across all utterances pre- intervention and post- intervention at the child level.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Hustad, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison Waisman Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months after publication of primary outcomes, and ending 5 years after that date.
Access Criteria: Data will be shared with researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose. Data will be shared for the following types of analyses: Independent verification of study outcomes or to conduct subsequent clinical research.
  Proposals should be directed to kchustad@wisc.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- [Background] Sakash A, Mahr TJ, Natzke PEM, Hustad KC. Effects of Rate Manipulation on Intelligibility in Children With Cerebral Palsy. Am J Speech Lang Pathol. 2020 Feb 7;29(1):127-141. doi: 10.1044/2019_AJSLP-19-0047. Epub 2019 Dec 23. PMID 31869242
- [Background] Korkalainen J, McCabe P, Smidt A, Morgan C. Motor Speech Interventions for Children With Cerebral Palsy: A Systematic Review. J Speech Lang Hear Res. 2023 Jan 12;66(1):110-125. doi: 10.1044/2022_JSLHR-22-00375. Epub 2023 Jan 9. PMID 36623233
- [Background] Levy ES, Chang YM, Ancelle JA, McAuliffe MJ. Acoustic and Perceptual Consequences of Speech Cues for Children With Dysarthria. J Speech Lang Hear Res. 2017 Jun 22;60(6S):1766-1779. doi: 10.1044/2017_JSLHR-S-16-0274. PMID 28655046
- [Background] Hustad KC, Lee J. Changes in speech production associated with alphabet supplementation. J Speech Lang Hear Res. 2008 Dec;51(6):1438-50. doi: 10.1044/1092-4388(2008/07-0185). Epub 2008 Jul 29. PMID 18664687
- [Background] Hustad KC, Jones T, Dailey S. Implementing speech supplementation strategies: effects on intelligibility and speech rate of individuals with chronic severe dysarthria. J Speech Lang Hear Res. 2003 Apr;46(2):462-74. PMID 14700386
- [Background] Stipancic KL, Yunusova Y, Berry JD, Green JR. Minimally Detectable Change and Minimal Clinically Important Difference of a Decline in Sentence Intelligibility and Speaking Rate for Individuals With Amyotrophic Lateral Sclerosis. J Speech Lang Hear Res. 2018 Nov 8;61(11):2757-2771. doi: 10.1044/2018_JSLHR-S-17-0366. PMID 30383220